CLINICAL TRIAL: NCT03406403
Title: A Comparative Study Between Laryngeal Mask Airway and Magensium Sulphate in Attenuating Systemic Stress Response During Emergence of Patients Undergoing Supratentorial Tumours.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Tarek Ahmed Radwan (Unknown); Mohamed Farid Mohamed (Unknown); Hamed Fathy Hamed (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-102-2017
Record Dates: First submitted 2017-12-26; First posted 2018-01-23 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: LMA Versus Mgso4 in Attenuating Stress Response During Emergence of Supratentorial Tumours Patients
MeSH Terms: interventions — Laryngeal Masks; Control Groups

STUDY DESIGN:
Intervention Model Description: We hypothesize that the LMA is more effective than Magnesium sulphate in attenuating systemic stress response during emergence of patients undergoing supratentorial tumours
Who Masked: Participant, Care Provider
Masking Description: The patients will be randomized into three equal groups. 60 slips of papers will be taken and labeled as group L (LMA), group M (Magnesium sulphate) and group C (Control). These slips will be placed in an envelope and one slip will be raised for each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Laryngeal mask airway group (Active Comparator): 20 slips of papers will be taken and labeled as group L (LMA) These slips will be placed in an envelope and one slip will be raised for each patient.
  Interventions: Device: Laryngeal mask airway; Drug: Magensium sulphate; Other: Control group (closure of anesthetics)
- Magensium sulphate group (Active Comparator): 20 slips of papers will be taken and labeled as group M (Mgso4) These slips will be placed in an envelope and one slip will be raised for each patient
  Interventions: Device: Laryngeal mask airway; Drug: Magensium sulphate; Other: Control group (closure of anesthetics)
- Control group (closure of anesthetics) (Active Comparator): 20 slips of papers will be taken and labeled as group C (Control) These slips will be placed in an envelope and one slip will be raised for each patient.
  Interventions: Device: Laryngeal mask airway; Drug: Magensium sulphate; Other: Control group (closure of anesthetics)

INTERVENTIONS:
Device: Laryngeal mask airway — After obtaining approval of the ethics committee of Kasr Al Ainy Hospitals and informed written consents from the patients, this study will be performed on 20 patients in Kasr Al Ainy Hospitals with ASA physical status I, II and ages between 18 and 60 years undergoing undergoing supratentorial tumours excision under general anesthesia
Drug: Magensium sulphate — After obtaining approval of the ethics committee of Kasr Al Ainy Hospitals and informed written consents from the patients, this study will be performed on 20 patients in Kasr Al Ainy Hospitals with ASA physical status I, II and ages between 18 and 60 years undergoing undergoing supratentorial tumours excision under general anesthesia
Other: Control group (closure of anesthetics) — After obtaining approval of the ethics committee of Kasr Al Ainy Hospitals and informed written consents from the patients, this study will be performed on 20 patients in Kasr Al Ainy Hospitals with ASA physical status I, II and ages between 18 and 60 years undergoing undergoing supratentorial tumours excision under general anesthesia

SUMMARY:
To evaluate the efficacy of replacement of ETT with LMA and administration of Magnesium sulphate at the end of the surgery in attenuating systemic stress response during emergence of patients undergoing supratentorial tumours

DETAILED DESCRIPTION:
Rapid recovery from neuroanesthesia and early neurological examination are desirable in most cases.(1)Although, Systemic and cerebral hemodynamic changes caused by extubation and emergence from anesthesia may endanger neurosurgical patients and increase the risk of postoperative intracranial hemorrhage and cerebral edema and may even result in the requirement of reoperation.(2) During this phase, heart rate and arterial blood pressure increase leading to increases in cerebral blood flow and intracranial pressure.(3) Some studies have reported such hemodynamic effects in up to 50% of patients after supratentorial craniotomy.(4,5) Replacing the endotracheal tube (ETT) with laryngeal mask airway (LMA) prior to emergence from anesthesia is safe and effectively reduces the cardiovascular response.(6) The potential protective benefit of this approach has not yet been demonstrated for awakening neurosurgery patients, however.

Magnesium is the forth most abundant cation in the body and the second most abundant intracellular cation. It activates many of the enzyme systems.(7) Magnesium sulphate inhibits catecholamines release from adrenergic nerve terminals and from adrenal medulla, through blocking N-type of Ca-channel at peripheral sympathetic nerve ending so it is used to decrease the adverse cardiovascular effects during larygeoscopy and endotracheal intubation.(8) But its role in attenuating stress response during extubation is not well studied and need more research.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I, II.
2. Ages between 18 and 60 years.
3. Body mass index (BMI) < 30.
4. Elective surgery

Exclusion Criteria:

1. Patients have cardiovascular, pulmonary, renal, hepatic and endocrine diseases.
2. Patients have any degree of disturbed conscious level.
3. Ages <18 or >60 years.
4. BMI >30.
5. Patients have history of allergy to Magnesium sulphate.
6. Patients have uncontrolled hypertension during preoperative assessment.
7. Patients have risk of aspiration (eg. hiatus hernia)
8. Patients have difficult airway management during intubation with direct laryngoscope or time of intubation >30 seconds.
9. Failed ventilation with LMA.
10. Emergency surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Mean arterial blood presure | 5 minutes from closure of anesthetics until 15 minutes after extubation
  Total dose of nitroglycerin needed in each group to maintain mean blood pressure within 20 % of basal line.

SECONDARY OUTCOMES:
Intracranial pressure Measurement | 1 and 10 minutes after extubation.
  Intracranial pressure will be measured at these moments: basal line preinduction, end of surgery, before extubation and 1, 10 minutes after extubation.
Quality of extubation | Time Onset of cough immediately after extubation
  Qualityof extubation will be evaluated based on cough immediately after extubation, using a five point rating scale
Level of consciousness | 5 and 15 minutes after extubation
  consciousness level will be recorded based on Ramasy score scale at 5 and 15 minutes after extubation, using the following indices
End of surgery and extubation | intraoperative
  Time interval between end of surgery and extubation in each group

CONTACTS AND LOCATIONS:
Overall Officials: Hamed Fathy, M.S, Principal Investigator — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Via scholar Gate